CLINICAL TRIAL: NCT00583271
Title: A Prospective Study of Endoscopic Ultrasound-guided Celiac (CB) Effectiveness
Brief Title: A Prospective Study of EUS Guided Celiac Block
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0205-04B; IRB #0205-04B
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Pancreatitis; Pancreatic Cancer
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatic Neoplasms | interventions — Triamcinolone; Triamcinolone Acetonide; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: subjects who are getting a celiac block for chronic pancreatitis
  Interventions: Drug: triamcinolone
- 2: subjects who are getting a celiac block for pancreatic cancer
  Interventions: Drug: 98% dehydrated alcohol

INTERVENTIONS:
Drug: triamcinolone — 80mg of triamcinolone injected into the celiac ganglion during the EUS-CB
  Other Names: Kenalog 80mg
  Groups: 1
Drug: 98% dehydrated alcohol — 10ml of 98% dehydrated alcohol injected into the celiac ganglion during the EUS-CB
  Groups: 2

SUMMARY:
The purpose of this prospective study is to measure the clinical effectiveness of EUS-guided CB in subjects, 50 who have chronic pancreatitis and 50 who have pancreatic cancer, that are already undergoing celiac block for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic abdominal pain from documented chronic pancreatitis or pancreatic cancer or other visceral malignancy that are undergoing EUS-guided CB (for purposes other than this study) will be eligible to participate in this study.
* Patients with chronic pancreatitis and pancreatic cancer must have documented disease by CT, ERCP, or EUS.
* No evidence of dementia or altered mental status that would prohibit the giving and understanding of informed consent, and no evidence of psychiatric risk that would preclude adequate compliance with this protocol.
* Patient must provide signed written informed consent

Exclusion Criteria:

* Patients that have had a previous celiac plexus block are eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with abdominal pain from documented chronic pancreatitis or pancreatic cancer that are referred for EUS-guided celiac block.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2002-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University
Locations (1):
- Clarian Health: Indiana University Hospital, Indianapolis, Indiana, United States